CLINICAL TRIAL: NCT02997033
Title: Longitudinal Extension Phase of Sibling Pair Linkage Analysis of Bone Mineral Density / Geometry and Sex Steroid and Thyroid Status in Healthy Young Men
Brief Title: SIBlos EXtension Study (SIBEX)
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Organization: University Hospital, Ghent (Other)
Other Study IDs: 2013/1090
Record Dates: First submitted 2016-12-14; First posted 2016-12-19 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Bone Density; Gonadal Steroid Hormones; Thyroid Hormones
Keywords: Bone; Sex steroids; Body composition; Men
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Venous blood sampling after overnight fast, with whole blood, serum and plasma samples to be retained
  * Second void urine samples to be retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Total study cohort
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Population-based, longitudinal cohort study designed to evaluate changes in bone mineral density, bone geometry, body composition, parameters reflecting muscle force, and sex steroid status in healthy young men, as well as their interactions, over a period of +-10 years.

DETAILED DESCRIPTION:
Osteoporosis is a common disorder affecting both sexes, with a lifetime risk of sustaining a fragility fracture at age 50 y estimated at 40-50% in women and 13-22% in men. The age-specific fracture risk in men is about half that in women, which results in part from the achievement of a higher bone mass in men, in particular of larger bone size during growth. Bone size, mass and strength in the elderly depend on the accrual and loss of bone through time. Not only from an epidemiological but also from a potentially preventive viewpoint, it is important to understand the determinants of the components and to identify risk and protective factors for bone accrual or loss through life.

Hormonal status in men, e.g. gonadal and thyroid hormone levels, has a wide range of effects on different body compartments. For both thyroid and gonadal steroid levels, there exists a wide inter-individual variation, even among healthy young men. Up till now, it is not clear whether this variation represents true differences in hormonal exposure or whether it represents an inter-individual variation in hormonal responsiveness. Since prevalence of both thyroid disorders and age- and obesity-associated hypogonadism is rather high, it is relevant to assess determinant and clinical correlates of the between-subject variation in sex steroid and thyroid hormone status.

Our research department therefore undertook a cross-sectional, population-based study in healthy men aged 25-45 years with the aim to investigate determinants of peak bone mass and between-subject variation in gonadal and thyroid hormone status (SIBLOS study). In total, 1114 men were recruited from 2002 till 2009. Herein, we focused on genetic determinants (SNPs, single nucleotide polymorphisms) contributing to between-subject differences in bone mass, as well as on the interrelationship between body composition, bone mass, density and size, lifestyle and hormonal status (sex steroids, thyroid hormones). In addition, we assessed determinants of sex steroid and thyroid hormone status, again focusing on genetic polymorphisms, body composition and lifestyle factors. The investigations in the SIBLOS study have been performed using state-of-the-art technology such as dual-energy X-ray absorptiometry and peripheral quantitative computed tomography for evaluating bone, muscle and body composition parameters; assessment of anthropometric parameters by well-trained personnel; validated questionnaires regarding lifestyle, physical activity and calcium intake; the use of liquid gas chromatography / mass spectrometry for assessing serum hormonal levels; using KASPar technology for genotyping after a high-yield DNA extraction procedure.

From this cross-sectional study, for example, following results have emerged:

* Estradiol seems to be the main sex steroid associated with bone mineral density and bone geometry, whereas testosterone was weakly associated with parameters reflecting muscle strength. In addition, serum estradiol levels might modulate the impact of physical activity on bone size at the tibia.
* Smokers presented with a higher prevalence of previous fractures, especially if they started smoking at younger age. This could be partly explained by the observation of lower bone mineral density and a thinner cortex in smokers.
* Physical activity, muscle mass and parameters reflecting muscle force are strongly associated with bone size; whereas fat mass displayed an inverse association with bone mass and size.
* Birth weight is associated with higher testosterone levels at adult age; in addition weight gain higher/lower than expected during life associated with lower/higher testosterone levels at adult age.
* Serum levels of sex-hormone binding globulin are positively associated with bone size in adult men.
* Higher serum thyroid hormone levels are associated with lower bone mineral density and cortical bone area.
* A less favorable body composition (higher fat and lower muscle mass) and insulin resistance are associated with higher serum thyroid hormone concentrations.
* Serum thyroid hormone levels are influenced by SNPs in the monocarboxylate transporter (MCT)-8 gene.
* Testosterone serum levels are associated with genetic polymorphisms in the genes encoding for the androgen receptor and sex-hormone binding globulin.

Our initial analyses in this SIBLOS population are cross-sectional. Although revealing, this, as any, cross-sectional study has limitations, mainly because the associations do not allow conclusions about direction nor causality. To add prospective elements to the acquired data and to investigate changes over time, we plan to perform a longitudinal follow-up in this study population (SIBEX - SIBlos EXtension study), and as in the mean time knowledge has increased and new questions have emerged, additional investigations are intended. The general aims of this follow-up study include the evaluation of changes in bone mineral density, bone geometry, body composition, parameters reflecting muscle force and sex steroid status in healthy young men, +-10 years after their initial evaluation in the SIBLOS cohort.

ELIGIBILITY:
Inclusion Criteria:

* Full participation in the first SIBLOS study
* Informed consent

Exclusion Criteria:

* Unwillingness or inability to participate
* Medication or disease known to affect bone metabolism, body composition and/or sex steroid metabolism:
* malignancy (previous or current)
* systemic diseases (auto-immune and rheumatoid pathology, ankylosing spondylitis)
* previous or current systemic use of glucocorticoids for more than 3 months, irrespective or dose
* use of glucocorticoid injections in previous 3 months
* use of inhalation glucocorticoids more than 500 µg / day
* previous or current thyroxin therapy (Graves disease, thyroidectomy)
* current insulin use for diabetes mellitus
* previous or current (anti-) androgen treatment or treated hypogonadism
* previous or current anti-epileptic drugs (phenytoin, valproate, carbamazepine, oxcarbazepine/carbamazepine, primidone)
* previous or current hyperthyroidism
* previous or current hyperparathyroidism or serum calcaemia < 8.5 or > 11 mg/dL
* hypocalcaemia (corrected for albumin, confirmed in 2 measurements)
* cystic fibrosis
* orchidectomy irrespective of underlying cause
* history of immobilisation > 3 months or immobilisation > 4 weeks within previous 6 months
* previous or current history of eating disorder
* serum creatinine > 2 mg% (estimated creatinine clearance < 35 mL/min)
* known diseases affecting growth, collagen, bone development or body composition (OI, otosclerosis, AIDS, ...)
* previous or current gastrointestinal malabsorption (gastrectomy, Crohn's disease, ulcerative colitis, coeliac disease, haemochromatosis)
* alcoholism (> 42 units per week)
* organ transplant recipients
* previous or current treatment for osteoporosis
* previous treatment for cryptorchidism irrespective of age
* current varicocoele or treatment for varicocoele after the age of 25 years (no exclusion if testosterone level in blood is normal)
* BMI > 42.3 kg/m²

Min Age: 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants of the first SIBLOS study (recruited between 2002 and 2009)
Sampling Method: Non-Probability Sample
Enrollment: 709 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in bone mineral density | ten years
  Change in bone mineral density vs. baseline (= study visit in SIBLOS study)

SECONDARY OUTCOMES:
Change in sex steroid levels | ten years
  Change in sex steroid levels vs. baseline (= study visit in SIBLOS study)
Change in body composition | ten years
  Change in body composition vs. baseline (= study visit in SIBLOS study)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Lapauw, M.D., Ph.D., Principal Investigator — University Ghent
Locations (1):
- Ghent University Hospital, Dept. of Endocrinology, Ghent, Belgium

REFERENCES:
- [Background] Kaptoge S, da Silva JA, Brixen K, Reid DM, Kroger H, Nielsen TL, Andersen M, Hagen C, Lorenc R, Boonen S, de Vernejoul MC, Stepan JJ, Adams J, Kaufman JM, Reeve J. Geographical variation in DXA bone mineral density in young European men and women. Results from the Network in Europe on Male Osteoporosis (NEMO) study. Bone. 2008 Aug;43(2):332-339. doi: 10.1016/j.bone.2008.04.001. Epub 2008 Apr 16. PMID 18519175
- [Background] Bogaert V, Taes Y, Konings P, Van Steen K, De Bacquer D, Goemaere S, Zmierczak H, Crabbe P, Kaufman JM. Heritability of blood concentrations of sex-steroids in relation to body composition in young adult male siblings. Clin Endocrinol (Oxf). 2008 Jul;69(1):129-35. doi: 10.1111/j.1365-2265.2008.03173.x. PMID 18598274
- [Background] Lapauw BM, Taes Y, Bogaert V, Vanbillemont G, Goemaere S, Zmierczak HG, De Bacquer D, Kaufman JM. Serum estradiol is associated with volumetric BMD and modulates the impact of physical activity on bone size at the age of peak bone mass: a study in healthy male siblings. J Bone Miner Res. 2009 Jun;24(6):1075-85. doi: 10.1359/jbmr.081260. PMID 19113912
- [Background] Vanbillemont G, Bogaert V, De Bacquer D, Lapauw B, Goemaere S, Toye K, Van Steen K, Taes Y, Kaufman JM. Polymorphisms of the SHBG gene contribute to the interindividual variation of sex steroid hormone blood levels in young, middle-aged and elderly men. Clin Endocrinol (Oxf). 2009 Feb;70(2):303-10. doi: 10.1111/j.1365-2265.2008.03365.x. Epub 2008 Aug 4. PMID 18681858
- [Background] Bogaert V, Vanbillemont G, Taes Y, De Bacquer D, Deschepper E, Van Steen K, Kaufman JM. Small effect of the androgen receptor gene GGN repeat polymorphism on serum testosterone levels in healthy men. Eur J Endocrinol. 2009 Jul;161(1):171-7. doi: 10.1530/EJE-09-0123. Epub 2009 Apr 21. PMID 19383805
- [Background] Taes YE, Lapauw B, Vanbillemont G, Bogaert V, De Bacquer D, Zmierczak H, Goemaere S, Kaufman JM. Fat mass is negatively associated with cortical bone size in young healthy male siblings. J Clin Endocrinol Metab. 2009 Jul;94(7):2325-31. doi: 10.1210/jc.2008-2501. Epub 2009 Apr 28. PMID 19401374
- [Background] Taes Y, Lapauw B, Vanbillemont G, Bogaert V, De Bacquer D, Goemaere S, Zmierczak H, Kaufman JM. Early smoking is associated with peak bone mass and prevalent fractures in young, healthy men. J Bone Miner Res. 2010 Feb;25(2):379-87. doi: 10.1359/jbmr.090809. PMID 19653814
- [Background] Vanbillemont G, Lapauw B, Bogaert V, De Naeyer H, De Bacquer D, Ruige J, Kaufman JM, Taes YE. Birth weight in relation to sex steroid status and body composition in young healthy male siblings. J Clin Endocrinol Metab. 2010 Apr;95(4):1587-94. doi: 10.1210/jc.2009-2149. Epub 2010 Feb 3. PMID 20130068
- [Background] Taes Y, Lapauw B, Griet V, De Bacquer D, Goemaere S, Zmierczak H, Kaufman JM. Prevalent fractures are related to cortical bone geometry in young healthy men at age of peak bone mass. J Bone Miner Res. 2010 Jun;25(6):1433-40. doi: 10.1002/jbmr.17. PMID 20200932
- [Background] Vanbillemont G, Lapauw B, Bogaert V, Goemaere S, Zmierczak HG, Taes Y, Kaufman JM. Sex hormone-binding globulin as an independent determinant of cortical bone status in men at the age of peak bone mass. J Clin Endocrinol Metab. 2010 Apr;95(4):1579-86. doi: 10.1210/jc.2009-2189. Epub 2010 Feb 4. PMID 20133463
- [Background] Roef G, Lapauw B, Goemaere S, Zmierczak H, Fiers T, Kaufman JM, Taes Y. Thyroid hormone status within the physiological range affects bone mass and density in healthy men at the age of peak bone mass. Eur J Endocrinol. 2011 Jun;164(6):1027-34. doi: 10.1530/EJE-10-1113. Epub 2011 Mar 10. PMID 21393448
- [Background] Vanbillemont G, Lapauw B, De Naeyer H, Roef G, Kaufman JM, Taes YE. Sex hormone-binding globulin at the crossroad of body composition, somatotropic axis and insulin/glucose homeostasis in young healthy men. Clin Endocrinol (Oxf). 2012 Jan;76(1):111-8. doi: 10.1111/j.1365-2265.2011.04155.x. PMID 21711374
- [Background] Boudin E, Piters E, Fransen E, Nielsen TL, Andersen M, Roef G, Taes Y, Brixen K, Van Hul W. Association study of common variants in the sFRP1 gene region and parameters of bone strength and body composition in two independent healthy Caucasian male cohorts. Mol Genet Metab. 2012 Mar;105(3):508-15. doi: 10.1016/j.ymgme.2011.11.189. Epub 2011 Nov 23. PMID 22178351
- [Background] Boudin E, Piters E, Nielsen TL, Andersen M, Roef G, Taes Y, Brixen K, Van Hul W. Single nucleotide polymorphisms in sFRP4 are associated with bone and body composition related parameters in Danish but not in Belgian men. Mol Genet Metab. 2012 Jul;106(3):366-74. doi: 10.1016/j.ymgme.2012.04.021. Epub 2012 May 2. PMID 22608881
- [Background] Roef G, Lapauw B, Goemaere S, Zmierczak HG, Toye K, Kaufman JM, Taes Y. Body composition and metabolic parameters are associated with variation in thyroid hormone levels among euthyroid young men. Eur J Endocrinol. 2012 Nov;167(5):719-26. doi: 10.1530/EJE-12-0447. Epub 2012 Sep 6. PMID 22956557
- [Background] Van Camp JK, Beckers S, Zegers D, Boudin E, Nielsen TL, Andersen M, Roef G, Taes Y, Brixen K, Van Hul W. Genetic association study of WNT10B polymorphisms with BMD and adiposity parameters in Danish and Belgian males. Endocrine. 2013 Aug;44(1):247-54. doi: 10.1007/s12020-012-9869-7. Epub 2013 Jan 17. PMID 23325361
- [Background] Roef GL, Rietzschel ER, De Meyer T, Bekaert S, De Buyzere ML, Van daele C, Toye K, Kaufman JM, Taes YE. Associations between single nucleotide polymorphisms in thyroid hormone transporter genes (MCT8, MCT10 and OATP1C1) and circulating thyroid hormones. Clin Chim Acta. 2013 Oct 21;425:227-32. doi: 10.1016/j.cca.2013.08.017. Epub 2013 Aug 24. PMID 23978482
- [Background] Roef G, Taes Y, Toye K, Goemaere S, Fiers T, Verstraete A, Kaufman JM. Heredity and lifestyle in the determination of between-subject variation in thyroid hormone levels in euthyroid men. Eur J Endocrinol. 2013 Oct 21;169(6):835-44. doi: 10.1530/EJE-13-0265. Print 2013 Dec. PMID 24086088
- [Background] De Naeyer H, Bogaert V, De Spaey A, Roef G, Vandewalle S, Derave W, Taes Y, Kaufman JM. Genetic variations in the androgen receptor are associated with steroid concentrations and anthropometrics but not with muscle mass in healthy young men. PLoS One. 2014 Jan 23;9(1):e86235. doi: 10.1371/journal.pone.0086235. eCollection 2014. PMID 24465978
- [Background] Gysel T, Calders P, Cambier D, Roman de Mettelinge T, Kaufman JM, Taes Y, Zmierczak HG, Goemaere S. Association between insulin resistance, lean mass and muscle torque/force in proximal versus distal body parts in healthy young men. J Musculoskelet Neuronal Interact. 2014 Mar;14(1):41-9. PMID 24583539
- [Background] Verroken C, Zmierczak HG, Goemaere S, Kaufman JM, Lapauw B. Association of Jumping Mechanography-Derived Indices of Muscle Function with Tibial Cortical Bone Geometry. Calcif Tissue Int. 2016 May;98(5):446-55. doi: 10.1007/s00223-015-0094-2. Epub 2015 Dec 16. PMID 26671019
- [Background] Verroken C, Zmierczak HG, Goemaere S, Kaufman JM, Lapauw B. Maternal age at childbirth is associated with offspring insulin sensitivity: a cross-sectional study in adult male siblings. Clin Endocrinol (Oxf). 2017 Jan;86(1):52-59. doi: 10.1111/cen.13253. Epub 2016 Nov 2. PMID 27726168
- [Derived] Verroken C, Zmierczak HG, Goemaere S, Kaufman JM, Lapauw B. Bone Turnover in Young Adult Men: Cross-Sectional Determinants and Associations With Prospectively Assessed Bone Loss. J Bone Miner Res. 2018 Feb;33(2):261-268. doi: 10.1002/jbmr.3303. Epub 2017 Nov 17. PMID 28987002